CLINICAL TRIAL: NCT05086094
Title: Intermediate-Size Patient Population Expanded Access Protocol of Verdiperstat in Patients With Multiple System Atrophy (MSA)
Brief Title: Expanded Access Protocol of Verdiperstat in Patients With Multiple System Atrophy (MSA)
Status: No longer available | Type: Expanded Access
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BHV3241-401
Record Dates: First submitted 2021-10-08; First posted 2021-10-20 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2021-10

CONDITIONS: Multiple System Atrophy (MSA)
Keywords: Multiple System Atrophy; MSA; verdiperstat; BHV3241; MPO inhibitor; Myeloperoxidase inhibitor; MSA-P; MSA-C
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: BHV3241, verdiperstat — BHV3241/Verdiperstat 600mg BID

SUMMARY:
The purpose of this expanded access program is to provide access to the investigational drug verdiperstat in patients with Multiple System Atrophy (MSA). Expanded access allows patients with a serious or a life-threatening disease or condition access to an investigational drug when no satisfactory approved treatment options are available.

ELIGIBILITY:
Inclusion Criteria:

1. with a diagnosis of probable or possible MSA documented by a physician according to consensus clinical criteria,5 including patients with MSA of either subtype, MSA-P or MSA-C.
2. able to swallow whole tablets without crushing or chewing.
3. with established care with a physician at the specialized MSA center involved in the protocol and will maintain this clinical care throughout the duration of the EAP.
4. not eligible for an ongoing clinical study with verdiperstat and/or an ongoing EAP for MSA

Exclusion Criteria:

1. Based on the Physician's judgement, any condition (including history of a clinically significant or unstable medical condition or lab abnormality) that would interfere with the patient's ability to comply with the EAP instructions, visit schedule, requirements and/or procedures, place the patient at unacceptable risk, or confound/interfere with the adequate assessment/interpretation of data; including difficulty swallowing verdiperstat tablets or any other sound medical, psychiatric and/or social reason.
2. Presence of clinically significant thyroid disease despite treatment and/or TSH >10 mIU/ L at Screening/Baseline, confirmed by repeat.
3. Patient is known to have acute or chronic liver disease that is clinically significant in the Prescriber's judgment
4. First or second dose of COVID-19 vaccination within 7 days of first dose of verdiperstat.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Morrisville, North Carolina, United States